CLINICAL TRIAL: NCT00999453
Title: The Effects of Lowering Low-density Lipoprotein Cholesterol Levels to New Targets on Cardiovascular Complications in Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Center for End Stage Renal Disease, Korea (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Shin-Wook Kang, Yonsei University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-02
Record Dates: First submitted 2009-10-18; First posted 2009-10-21 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2009-10

CONDITIONS: Hypercholesterolemia
Keywords: LDL-cholesterol; Prevalent peritoneal dialysis patients with hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Cholesterol, LDL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LDL-cholesterol 70 mg/dL or lower (Experimental): 'Experimental arm' is defined as patients treated to lower the level of low-density lipoprotein to 70 mg/dl or lower. 'Control arm' is defined as patients treated to lower low-density lipoprotein to a level of 100 mg/dl or lower.
  Interventions: Other: LDL-cholesterol
- LDL-cholesterol 100 mg/dL or lower (Active Comparator): 'Experimental arm' is defined as patients treated to lower the level of low-density lipoprotein to 70 mg/dl or lower. 'Control arm' is defined as patients treated to lower low-density lipoprotein to a level of 100 mg/dl or lower.
  Interventions: Other: LDL-cholesterol

INTERVENTIONS:
Other: LDL-cholesterol — This is a 2-arm, open label, multi-center, randomized trial comparing aggressive to standard treatment of LDL-cholesterol. After screening, randomization, participants will be seen every 3 months during the follow-up period. An LDL-cholesterol 100 mg/dL is the goal for the standard group and the target for the aggressive group is 70 mg/dL. A lipid lowering algorithm has been developed based on the NCEP-ATP III recommendation which is used as a general guideline, allowing alterations based on the individual participants needs.

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality in dialysis patients. Although significant improvements have been made in the management of CVD in the general population, it is not known whether these interventions would result in similar benefits in end stage renal disease patients.

Clinical studies conducted in the general population and in patients with established cardiovascular disease have found a strong independent association between lipid lowering, primarily LDL-cholesterol, and the risk of all-cause and cardiovascular mortality.

Therefore the National Cholesterol Education Panel (NCEP) has provided guidelines to lower LDL cholesterol levels to a goal of ≤100 mg/dl in patients with major risk factors of coronary heart disease. Moreover, the recent Adult Treatment Panel III (ATP III) guidelines provide an option to lower LDL cholesterol levels to a goal of <70 mg/dl in patients with very high risks for coronary heart disease.

The National Kidney Foundation K/DOQI guideline regards dialysis patients as having high risks for coronary heart disease and consequently recommends the LDL cholesterol level to be maintained under 100 mg/dl. This recommendation is in parallel to the NCEP ATP III guideline which has been proposed for the general population. However, data regarding cholesterol levels in dialysis patients have been conflicting, with some observational studies demonstrating and some not demonstrating a clear, relationship between LDL and cardiovascular end-points. In addition few randomized studies have been conducted in CKD patients.

An observational retrospective analysis of patients receiving hemodialysis, the U.S. Renal Data System Morbidity and Mortality Study, showed that the risk for cardiovascular mortality was decreased by 36 percent among patients receiving statins, compared to those who did not. Whereas, a most recent large prospective study in diabetic hemodialysis patients failed to demonstrate a significant reduction in cardiovascular endpoints with statin therapy.

Moreover, although HD and PD patients both develop chronic hypervolemia and inflammation as common findings, the relationship between risk factors and outcome may differ between these two treatment methods. The likely role of glucose from the dialysate in causing dyslipidemia in PD patients inherits a different strength of association between cholesterol level and outcome in HD and PD patients.

Therefore, this study aims to examine the clinical outcomes of treating chronic peritoneal dialysis patients with dyslipidemia to lower cholesterol levels, randomly assigning patients to either aggressive targets of LDL cholesterol of 70 mg/dl or current standard targets of LDLD cholesterol of 100 mg/dl.

ELIGIBILITY:
Inclusion criteria:

1. End-stage renal disease patients treated with peritoneal dialysis for 3 or more months
2. LDL cholesterol 100 mg/dl or higher within 3 months and total cholesterol level 220 mg/dl or higher

Exclusion criteria:

1. Hypersensitivity to statin, ezetimibe, fenofibrate
2. Acute MI, angina, cerebrovascular accident, vascular intervention within the last 6 months
3. Chronic obstructive pulmonary disease
4. alanine transaminase > 3 times the upper normal limit
5. creatine kinase > 3 times the upper normal limit
6. Patients suffering form non-cardiac diseases with estimated survival less than 2 years
7. Inevitable of cyclosporin, warfarin use
8. Currently pregnant or breast feeding
9. Any condition that might limit long-term compliance (e.g., psychiatric disorders)
10. Participation in another clinical trial within 30 days prior to enrollment

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Cardiovascular complication including acute coronary syndrome, cerebrovascular infarction and cardiovascular death | 5 years (after detecting Cardiovascular complication)

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Wook Kang, M.D., PhD., Principal Investigator — professor of division of Nephrology, Severance Hospital, Korea
Locations (2):
- South Korea (2):
  - Kyungpook National University Hospital, Daegu
  - Severance Hospital, Seoul